CLINICAL TRIAL: NCT05566522
Title: Development of a Comprehensive Kinesiophobia Rating Scale
Brief Title: Comprehensive Kinesiophobia Rating Scale
Status: Completed | Type: Observational
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Burcu Talu, assoc. prof., Inonu University
Other Study IDs: 2021/1781
Record Dates: First submitted 2022-09-30; First posted 2022-10-04 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2022-07

CONDITIONS: Kinesiophobia; Movement Phobia
Keywords: kinesiophobia; scale; movement
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Those between the ages of 20-75, Those with musculuskeletal disorders, choronic and neurological disease
- Control Group: Healty group

SUMMARY:
The aim of this study is to comprehensively evaluate the fear of movement in different diseases. Individuals between the ages of 20-75 will be included in the study. Survey development phase; It consisted of literature review, qualitative research and the creation of the draft form. The literature review includes the creation of an item pool through a detailed examination of the studies on scales assessing kinesiophobia and the questionnaires used. Scale Postural control, balance, pain, anxiety/depression, 5' likert type orientation with 28 items consisting of sensory and interaction. 0 strongly disagree, 1: disagree, 2: not sure, 3: have, 4: have. Each section's own score and total score will be calculated out of 100. TAMPA Kinesiophobia Scale will be used to calculate the convergent validity of the questionnaire.

DETAILED DESCRIPTION:
The aim of this study is to comprehensively evaluate the fear of movement in different diseases. Individuals between the ages of 20-75, those with musculoskeletal, and chronic diseases, individuals with a Standard Mini-Mental Test Score of 24 above, individuals who voluntarily agreed to participate in the study, and individuals with informed consent will be included in the study. Individuals with cardiac and pulmonary problems that may hinder the study, individuals who do not allow mental assessment, individuals who cannot read and write in Turkish and who cannot answer the questions will not be included in the study. The deductive/inductive method will be used to create the survey questions. Survey development phase; It was composed of literature review, qualitative research, and the creation of the draft form. The literature review includes the creation of an item pool through a detailed examination of the studies on scales evaluating kinesiophobia and the questionnaires used. The draft created as a result of the literature review was sent to the linguist, who evaluated the subject in terms of meaning and grammar. Then, 10 expert opinions were asked to rate each question in terms of relevance, clarity, simplicity, and specificity, and were determined as inappropriate, somewhat appropriate, highly relevant, and very appropriate. Then, a pilot application will be made to evaluate the face validity of the questionnaire. At this stage, the pilot study of the scale, which has passed the expert opinion, will be carried out with a small sample. The scale was created in a 5-point Likert type format with 28 items consisting of Postural control/balance, pain, anxiety/depression, sensory and social interaction sections. 0 strongly disagree, 1: disagree, 2: not sure, 3: agree, 4: completely agree. The score of each section and the total score will be calculated out of 100. Then, criterion-based validity (concurrent validity) method will be used to evaluate the validity of the questionnaire, and at this stage, individuals will be determined from the relevant population by non-probabilistic sampling method; Groups will be assigned with the stratified sampling method. In the other stage, TAMPA Kinesiophobia Scale will be used to determine the convergent validity of the questionnaire. At the last stage, the reliability of the questionnaire will be evaluated. Its reliability will be evaluated by the test-retest method. The scale will be administered on the same subjects at two different times (1-3 days apart) under the same conditions. In our double-blind randomized study, Inter-observer Consistency will be tested by using Correlation - Kendall's Coefficient of Concordance to calculate the agreement between independent observers. The same procedures will be done for the healthy individuals in the control group. The control group will also be selected from the relevant population with an improbable random method. The Cronbach Alpha Reliability Coefficient will be used to evaluate the internal consistency of the study.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 20-75,
* Those with musculoskeletal disorders,
* Those with neurological disorders,
* Those with chronic illness,
* Individuals who correctly answered all orientation questions in the Standard Mini Mental Test,
* Individuals who agree to participate in the study voluntarily,
* Individuals with informed consent will be included in the study

Exclusion Criteria:

* Individuals with cardiac and pulmonary problems that may interfere with the study,
* Individuals who cannot cooperate,
* Individuals who are illiterate in Turkish and cannot answer questions Exclusion criteria of volunteers
* Individuals who could not adapt to the parameters during the evaluation,
* Individuals who want to leave the study voluntarily

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who will voluntarily participate in the study will be evaluated through the online platform.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2023-02-22 (Actual)

PRIMARY OUTCOMES:
Kinesiophobia Assesment | 5 mounts
  Tampa Kinesiophobia Scale will use in this study. The Tampa Kinesiophobia Scale (TKS) is one of them, and it's commonly used in the literature to assess kinesiophobia. It has 17 questions designed to assess fear of moving.
Kinesiophobia Assesment | 5 mounts
  It will be evaluated with the comprehensive kinesiophobia rating scale that we aim to develop.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Talu, Assoc. Prof, Study Director — Inonu University; Havva Adlı, PhD. (cand)., Principal Investigator — Inonu University; Gülfem Ezgi ÖZALTIN, PhD. (cand), Principal Investigator — Inonu University
Locations (1):
- Inonu University, Malatya, Turkey (Türkiye)